CLINICAL TRIAL: NCT05343325
Title: Neoadjuvant Low-dose Radiotherapy, Tislelizumab, Combined With Albumin-bound Paclitaxel and Cisplatin in Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma (NeoRTPC02): an Open Label, Single-arm, Phase II Clinical Trial
Brief Title: The Efficacy and Safety of Neoadjuvant Low-dose Radiotherapy Combined With Chemoimmunotherapy in Locally Advanced HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Dongguan People's Hospital (Other Government)
Responsible Party: Principal Investigator, Zhigang Liu, Director, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.ZLZX.011
Record Dates: First submitted 2022-04-13; First posted 2022-04-25 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Neoadjuvant Treatment
Keywords: locally advanced HNSCC; neoadjuvant treatment; low-dose radiotherapy; pathological response rates
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab; Albumin-Bound Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose Radiotherapy, Tislelizumab, Combined With Albumin-bound Paclitaxel and Cisplatin (Experimental): Neoadjuvant therapy will be performed for a total of 2 cycles, with 21 days as a cycle, which includes: ① Low-dose radiotherapy: 1GY/1F, D1, D2, D8, D15, Q3W for two cycles, and the total dose of radiation in the two cycles will be GTV 8 Gy/8 F and GTVnd 8 Gy/8 F; ② Teilizumab: 200 mg D1, Q3W for two cycles; ③ Albumin-bound paclitaxel: 100mg/m2, D1, D8, D15, Q3W for two cycles; ④Cisplatin: 25mg/m2, D1, D8, D15, Q3W for two cycles.
  Interventions: Drug: Tislelizumab; Radiation: Low-dose radiotherapy

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab: 200 mg D1, Q3W for two cycles. Albumin-bound paclitaxel: 100mg/m2, D1, D8, D15, Q3W for two cycles. Cisplatin: 25mg/m2, D1, D8, D15, Q3W for two cycles.
  Other Names: Albumin-bound paclitaxel; Cisplatin
Radiation: Low-dose radiotherapy — Low-dose radiotherapy: 1GY/1F, D1, D2, D8, D15, Q3W for two cycles. The total radiation dose will be GTV 8Gy/8F, GTVnd 8 Gy/8F.

SUMMARY:
This is an open-label, single-arm, phase II clinical trial to explore the efficacy and safety of neoadjuvant low-dose radiotherapy combined with chemoimmunotherapy in resectable locally advanced head and neck squamous cell carcinoma. The eligible patients are scheduled to administered neoadjuvant low-dose radiotherapy, tislelizumab, combined with albumin-bound paclitaxel and cisplatin for two cycles. Radical resection will be performed in 3-4 weeks after two cycles of neoadjuvant therapy. The overall primary study hypothesis is that the novel neoadjuvant combination regime improves the pathological complete response (pCR) rate, with tolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated, histologically confirmed head and neck squamous cell carcinoma (oral cavity, oropharynx, hypopharynx or larynx), staging T3-4N0M0 or T1-4N1-3M0, III-IVB, according to the eighth edition of the AJCC staging system;
2. Eligible for radical surgery, as judged by surgeons.
3. Aged ≥ 18 years and ≤ 70 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
5. Life expectancy of more than 6 months.
6. At least one measurable lesion according to RECIST 1.1.
7. Adequate organ function, based on meeting all of the following criteria (no blood components and cytologic growth factors were received within 14 days prior to the test):

   1. Hemoglobin ≥ 90 g/L; absolute neutrophil count ≥ 1.5 × 109/L; and platelet count ≥ 100 × 109/L;
   2. Serum albumin ≥ 28 g/L;
   3. Total bilirubin ≤ 1.5 × upper limit of normal (ULN); ALT and AST ≤ 2.5 × ULN;
   4. Serum creatinine ≤ 1.5 × ULN and creatinine clearance rate ≥ 50 mL/min;
   5. Activated partial clotting enzyme time and international standardized ratio (INR) ≤ 1.5 × ULN (Patients on stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin with INR within the expected treatment range of anticoagulants can be screened ).

      43/5000
   6. Thyroid Stimulating Hormone (TSH) ≤ULN; If abnormal, T3 and T4 levels should be examined, and patients with normal T3 and T4 levels can be screened.
8. Women of childbearing age should agree to the use of contraception (e.g., intrauterine devices, birth control pills, or condoms) during drug administration and for 3 months thereafter.
9. Subjects voluntarily join the study and sign an informed consent form, with good compliance.

Exclusion Criteria (Patients will be excluded if any of the following criteria is met):

1. Pregnant or lactating women.
2. A history of allergies to PD-1 inhibitors or any of albumin-bound paclitaxel or cisplatin.
3. A history of other malignant tumors within the previous 5 years or at the time of enrollment, except for cured skin basal cell carcinoma and cervical in situ cancer, as well as thyroid papilloma.
4. Uncontrolled cardiac clinical symptoms or diseases, such as :(1) NYHA class II or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, and (4) patients with clinically significant ventricular or ventricular arrhythmias requiring intervention.
5. Have received any of the following treatments:

   1. Any research drug received prior to the first dose of the current research drug.
   2. Joined another clinical study at the same time, unless it is an observational (noninterventional) clinical study or an intervention during a follow-up.
   3. Needed systemic treatment with corticosteroids (more than 10 mg of prednisone or equivalent per day) or other immunosuppressants within 2 weeks prior to the first dose of the study drug, except for the use of corticosteroids for local inflammation and prevention of allergies or nausea and vomiting. In the absence of active autoimmune diseases, inhalation or partial use of steroids and adrenal corticosteroid replacements at doses greater than 10 mg per day of fentanyl equivalent is permitted.
   4. Live vaccines were administered within 4 weeks prior to the first administration of research drugs.
   5. Major surgery or severe trauma within four weeks of initial use of the study drug.
6. Serious infections (greater than grade 2 according to the Common Terminology Criteria for Adverse Events), such as severe pneumonia, bacteremia, and infection comorbidities, which required hospitalization, occurred within 4 weeks prior to the first dose of the study drug; baseline chest imaging examinations indicate the presence of active lung inflammation or symptoms and signs of infection within 2 weeks prior to the first dose of the study drug or indicate the need for oral or intravenous antibiotic treatment (excluding the use of preventive antibiotics).
7. A history of active autoimmune diseases and syndromes (including, but not limited to, interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, and hypothyroidism). Patients with vitiligo or cured childhood asthma/allergies that do not require any intervention in adulthood are not excluded.
8. A history of immunodeficiency, including HIV-positive status or other acquired congenital immunodeficiency diseases, or a history of organ transplantation and bone marrow transplantation.
9. Patients with active tuberculosis infection found by history or CT examination, or patients with active tuberculosis infection history within 1 year prior to enrollment, or patients with active tuberculosis infection history before 1 year without formal treatment.
10. Active hepatitis B (HBV DNA ≥ 2,000 IU/mL or 10,000 copies/mL) or hepatitis C (positive HCV antibody test and HCV RNA above the lower limit of detection).
11. Known history of psychotropic drug abuse, alcoholism and drug use.
12. Not suitable for inclusion, as judged by the researcher.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | 1 week after surgery
  the proportion of patients with no residual viable tumor cell under microscope

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | 1 week after surgery
  the proportion of patients with the percentage of residual viable tumor cells in the tumor bed less than 10%
Objective Response Rate (ORR) | 3-4 weeks after two cycles of neoadjuvant therapy
  the proportion of patients with radiographic objective responses (complete response and partial response)
Incidence of treatment-related adverse events | from the first day of treatment to 30 days after surgery
  CTCAE 5.0
Non-surgery-delay rate | 8 weeks after two cycles of neoadjuvant therapy
  the proportion of patients with surgical operation conducted more than four weeks longer than scheduled
EORTC QLQ-C30 | from 1 week before treatment to 30 days after surgery
  Quality of life evaluation
EORTC HN35 | from 1 week before treatment to 30 days after surgery
  Quality of life evaluation

OTHER OUTCOMES:
Progression-free survival (PFS) | from the first day of treatment to the follow up of 3 years
  3-year progression free survival rate
Overall survival (OS) | from the first day of treatment to the follow up of 3 years
  3-year overall survival rate

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Zhigang Liu, Dongguan

IPD SHARING:
Plan to Share IPD: No